CLINICAL TRIAL: NCT06638489
Title: Effects of High Intensity Focused Electromagnetic Therapy With Pelvic Floor Muscle Training on Urine Leakage and Quality of Life in Primipara or Multipara Women With Stress Urinary Incontinence: A Pilot for Randomised Controlled Trial
Brief Title: Effects of High Intensity Focused Electromagnetic Therapy With Pelvic Floor Muscle Training on Urine Leakage and Quality of Life in Primipara or Multipara Women With Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, LIU FANG, Principal Investigator, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N&HS00004
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group received both High-Intensity-Focused-Electromagnetic-Therapy (HIFEM) combined with Pelvic-Floor-Muscle-Training (PFMT)
  Interventions: Other: High-Intensity-Focused-Electromagnetic-Therapy (HIFEM); Other: Pelvic-Floor-Muscle-Training (PFMT)
- control group (Experimental): the control group received only Pelvic-Floor-Muscle-Training (PFMT)
  Interventions: Other: Pelvic-Floor-Muscle-Training (PFMT)

INTERVENTIONS:
Other: High-Intensity-Focused-Electromagnetic-Therapy (HIFEM) — The HIFEM stimulation was administered using an Emsella instrument (manufactured by BTL Industry Inc., Boston, MA). The frequency ranged between 50 and 60Hz, and the intensity was as high as the patient could tolerate, which was usually up to 100%.
  Arms: experimental group
Other: Pelvic-Floor-Muscle-Training (PFMT) — The PFMT protocol was that outlined by previous study. The participants were instructed to execute 5 rapid contractions over a span of 3 seconds and 10 prolonged contractions, each lasting between 3 to 8 seconds, with intervals of 10 seconds for relaxation in between, all while in a crook-lying position.

SUMMARY:
This study aimed to evaluate the impact of High-Intensity Focused Electromagnetic Therapy (HIFEM) combined with Pelvic Floor Muscle Training (PFMT) versus PFMT alone on urine leakage and quality of life in primiparous and multiparous women with stress urinary incontinence. Women aged 30 years or older exhibiting symptoms of stress urinary incontinence were randomized into two treatment groups. The experimental group received both HIFEM and PFMT, while the control group received only PFMT. The treatment continued for 6 weeks. Evaluations measured at baseline and post-intervention included the 1-hour Pad Test, the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI-SF), and sonography to assess bladder neck movement.

ELIGIBILITY:
Inclusion Criteria:

* Primipara or Multipara women aged 30 years or older with symptoms of stress urinary incontinence;

Exclusion Criteria:

* Those who had any contraindication for High-Intensity-Focused-Electromagnetic-Therapy (HIFEM);
* prior surgery for incontinence;
* taking drugs for bladder dysfunction or diuretics;
* hormone therapy;
* urgent or mixed urinary incontinence;
* incontinence associated with a neurologic condition;
* inability to perform voluntary pelvic floor muscle contractions;
* cognitive impairment or dementia, major neurological disorders (such as stroke, cerebral palsy, multiple sclerosis);
* inability to carry out the treatment or evaluation;
* uncontrolled hypertension.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
1-hour pad test | Baseline and the end of the 6-week intervention
  It measures the total amount of urine leakage by weighing the pad after performing several standardized activities over the course of an hour.

SECONDARY OUTCOMES:
International Consultation on Urinary Incontinence questionnaire (ICIQ-UI-SF) | Baseline and the end of the 6-week intervention
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI-SF) is a widely used tool designed to assess the severity and impact of urinary incontinence on an individual's quality of life. The scores from these items provide an overall score that ranges from 0 to 20, with higher scores indicating greater severity of urinary incontinence and a more significant impact on quality of life.
Bladder neck movement | Baseline and the end of the 6-week intervention
  The bladder neck movement was measured by sonography. The ultrasound scanner was a Clarius C3 HD3 (Clarius Mobile Health, Vancouver, Canada).

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Chan WS, Chow WT, Poon YT, Tsang CSL, Yuen HHL, Lui EWY, Wong YT, Tsang WWN. Effects of High-Intensity Focused Electromagnetic Therapy (HIFEM) With Pelvic Floor Muscle Training in Mothers Living With Incontinence: A Pilot for a Randomized Controlled Trial. Womens Health Issues. 2026 Jan 24:S1049-3867(25)00160-4. doi: 10.1016/j.whi.2025.12.002. Online ahead of print. PMID 41582071

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT06638489/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT06638489/ICF_001.pdf